CLINICAL TRIAL: NCT06169566
Title: Analysis of Gut Microbiome in Thai Women With Polycystic Ovary Syndrome and the Synbiotics Effect on Reproductive and Cardiovascular Risk: A Randomized Controlled Trial
Brief Title: The Synbiotics Effects in Polycystic Ovary Syndrome: A Randomized Controlled Trial
Acronym: PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maharaj Nakorn Chiang Mai Hospital (Other)
Responsible Party: Principal Investigator, Ploywarong Rueangket, MD., Maharaj Nakorn Chiang Mai Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OBG-2566-0568
Record Dates: First submitted 2023-11-27; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: PCOS- Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): synbiotics
  Interventions: Dietary Supplement: synbiotics
- non-intervention (Placebo Comparator): placebo
  Interventions: Combination Product: placebo

INTERVENTIONS:
Dietary Supplement: synbiotics — synbiotics
  Arms: Intervention
Combination Product: placebo — placebo
  Arms: non-intervention

SUMMARY:
The goal of this clinical trial is to compare the effect of synbiotics and placebo in Thai women with polycystic ovary syndrome. The main questions it aims to answer are:

* Do synbiotics have a positive effect on the gut microbiome?
* Do synbiotics have a positive effect on reproductive outcomes?
* Do synbiotics have a positive effect on cardiovascular outcomes? Participants will be randomized, and blinded to receive either synbiotics or placebo.

While placebo is a comparison group: Researchers will compare with placebo to see if the effects on reproductive and cardiovascular risk differ.

DETAILED DESCRIPTION:
Analysis of gut microbiome in Thai women with polycystic ovary syndrome and the synbiotics effect on reproductive and cardiovascular risk: A randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

- PCOS

Exclusion Criteria:

* ATB use

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome in polycystic ovary syndrome | 12 months
  Gut microbiome will be evaluated by metagenomic analysis of the stool exam of PCOS patient before and after receive synbiotics

SECONDARY OUTCOMES:
synbiotics effect on reproductive and cardiovascular risk | 12 months
  evaluation of the reproductive clinical (menstrual regularity, polycystic ovarian morphology on the ultrasound) and serum marker of cardiovascular risk (Lipid profile, HbA1C, fasting blood glucose, hsCRP) will be evaluated compare between synbiotics and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Ploywarong Rueangket, MD, Principal Investigator — Department of obstetrics and gynecoloy
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No